CLINICAL TRIAL: NCT00005969
Title: Phase II Study of ATRAGEN (Liposomal Tretinoin) in Patients With Relapsed or Refractory Hodgkin's Disease
Brief Title: Liposomal Tretinoin in Treating Patients With Recurrent or Refractory Hodgkin's Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study withdrawn.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID99-255; P30CA016672 (NIH); MDA-ID-99255 (Other: UT MD Anderson Cancer Center); NCI-103; CDR0000067952 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2000-07-05; First posted 2004-04-28 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Recurrence | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Liposomal Tretinoin (Experimental): Liposome by vein (IV) over 30 minutes every other day for 28 days and Chemotherapy.
  Interventions: Drug: Chemotherapy; Drug: Tretinoin Liposome

INTERVENTIONS:
Drug: Chemotherapy
Drug: Tretinoin Liposome — Liposome by vein (IV) over 30 minutes every other day for 28 days
  Other Names: ATRAGEN

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of liposomal tretinoin in treating patients who have recurrent or refractory Hodgkin's disease.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate, failure free survival, and progression free survival of patients with recurrent or refractory Hodgkin's disease treated with tretinoin liposome. II. Determine the toxicities of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to prior response to treatment (refractory vs recurrent vs post marrow transplant). Patients receive tretinoin liposome IV over 30 minutes every other day for 28 days. Treatment continues every 28 days for a total of 6 courses in the absence of disease progression or unacceptable toxicity. Patients who are eligible for stem cell or marrow transplant receive at least 2 courses before crossing over to transplant. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 105 patients (35 per strata) will be accrued for this study over 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent or refractory Hodgkin's disease Recurrent after partial or complete response after initial therapy OR Refractory after no response or progression after initial therapy At least 2 prior treatment regimens (radiotherapy considered separate if not part of planned combined modality) Bidimensionally measurable disease No active CNS disease

PATIENT CHARACTERISTICS: Age: 12 and over Performance status: Zubrod 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 500/mm3 Platelet count at least 20,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGPT less than 4 times upper limit of normal Renal: Creatinine no greater than 3.0 mg/dL Other: Not pregnant or nursing Fertile patients must use effective contraception Must not be eligible or willing to undergo treatment of a higher priority HIV negative No other prior malignancies within the last 5 years except basal cell carcinoma of the skin or carcinoma in situ of the cervix treated with curative intent No other concurrent serious illness or active infection No mental or social reasons that may preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: No more than 1 prior autologous stem cell or marrow transplant No prior allogenic stem cell or marrow transplant Chemotherapy: See Disease Characteristics Must be recovered from last regimen No prior retinoids, including tretinoin Endocrine therapy: No concurrent steroids Radiotherapy: See Disease Characteristics Must be recovered from last regimen Surgery: Not specified

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1999-09; Primary Completion 2001-01 (Actual)

PRIMARY OUTCOMES:
Patient Response Rate | 28 Day Cycles

CONTACTS AND LOCATIONS:
Overall Officials: Andreas H. Sarris, MD, PhD, Study Chair — M.D. Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org